CLINICAL TRIAL: NCT00324610
Title: Phase I/II Study of Tolerance and Pharmacokinetics With Capecitabine Given 5 Days Out of 7 in Metastatic Breast Cancer
Brief Title: Tolerance and Pharmacokinetics With Capecitabine 5 Out of 7 Days Regimen
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Pour La Recherche des Thérapeutiques Innovantes en Cancérologie (Other)
Other Study IDs: CAP 5/7; ARTIC / CAP 5/7
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2006-05-18 (Estimated); Status verified 2006-05

CONDITIONS: Breast Neoplasms; Chemotherapy
Keywords: fluoropyrimidines; metastases; pharmacokinetics; phase 1-2 study
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Capecitabine

INTERVENTIONS:
Drug: capecitabine

SUMMARY:
Standard administration of capecitabine use a 14 days administration. Routine practice in several intitution leads to use a 5 out of 7 days regimen, with less toxicity.

Purpose : to compare the pharmacokinetics of capecitabine, administered 5 days out of 7, as compared to the standard administration (14 days out of 21). The second end point is to compare toxicity with either regimen.

Method : Randomized study with two groups : one with standard administration , the second with 5/7 days regimen

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven breast adenocarcinoma
* Evaluable or measurable metastases
* HER-2 status 0 or 1 in immnohistochimy or negative in FISH/CISH
* Previously treated with anthracyclines and taxanes
* Age > = 18 y
* No more than two previous chemotherapy regimens for metastases
* No nervous central system involvement
* Hormonal therapy must have been stopped two weeks before enrollment
* Adequate biologic function
* Performance status OMS < = 2
* Signed informed consent

Exclusion Criteria:

* History of other malignancies, except basocellular cancer, in situ cervix carcinoma
* Gastro intestinal disease that might affect absorption of capecitabine
* Cardiac failure or angina pectoris uncontrolled
* Hypersensitivity for capecitabine, fluorouracil, or one of their excipient
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Concomitant anticancer therapy (included hormonotherapy)
* Concomitant radiotherapy
* Treatment with sorivudine and analogs
* Pregnant or breast feeding patients. Contraception methods excluding hormonal treatment is required.
* Inclusion in an experimental protocol within 30 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46
Dates: Start 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: eric levy, MD, Principal Investigator — HEGP , PARIS; joseph Gligorov, MD, Study Chair — HOPITAL TENON, PARIS; Michèle TUBIANA HULIN, MD, Study Chair — CENTRE RENE HUGUENIN, SAINT CLOUD, FRANCE; VERONIQUE DIERAS, MD, Study Chair — INSTITUT CURIE, PARIS france; Rémi LARGILLIER, MD, Study Chair — centre antoine lacassagne, NICE, France
Locations (1):
- Ho¨Pital Europeen Georges Pompidou, Paris, France